CLINICAL TRIAL: NCT00091559
Title: Phase IIb Multicenter Clinical Trial of Oral Suberoylanilide Hydroxamic Acid (SAHA) in Advanced Cutaneous T-cell Lymphoma
Brief Title: Oral SAHA (Suberoylanilide Hydroxamic Acid) in Advanced Cutaneous T-cell Lymphoma (0683-001)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0683-001; 2004_015
Record Dates: First submitted 2004-09-10; First posted 2004-09-14 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Cutaneous T-cell Lymphoma; Sezary Syndrome; Mycosis Fungoides
Keywords: CTCL
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Sezary Syndrome; Mycosis Fungoides | interventions — Vorinostat; Duration of Therapy

INTERVENTIONS:
Drug: MK0683, vorinostat, Suberoylanilide Hydroxamic Acid (SAHA) / Duration of Treatment 6 Months

SUMMARY:
A study for patients diagnosed with advanced cutaneous T-cell lymphoma (stage 1B or higher) who have progressive, persistent, or recurrent disease on or following 2 other therapies, one of which must have contained Targretin (bexarotene)or for patients who are not candidates or could not tolerate Targretin therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Cutaneous T-cell Lymphoma (Stage 1B or higher)
* Age: over 18 years of age
* Have the ability to swallow capsules.
* You must be at least 3 weeks from any prior chemotherapy or anticancer therapy treatment and have recovered from any side effects of that treatment.
* Patients also require adequate heart, liver, and kidney function.

Exclusion Criteria:

* Pregnant and nursing women and those with known allergy to the study drug are excluded from this study.
* Patients are excluded if they are currently receiving chemotherapy, radiation therapy, or other investigational anti-cancer therapy.
* Patients diagnosed with HIV, active hepatitis or who require intravenous antibiotics or antifungal agents are not permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2005-02-03 (Actual); Primary Completion 2005-11-23 (Actual); Study Completion 2006-03-13 (Actual)

PRIMARY OUTCOMES:
Objective response rate in patients with progressive, persistent, or recurrent disease.

SECONDARY OUTCOMES:
Response duration, relief of pruritis, time to progression, time to objective response, safety & tolerability in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Olsen EA, Kim YH, Kuzel TM, Pacheco TR, Foss FM, Parker S, Frankel SR, Chen C, Ricker JL, Arduino JM, Duvic M. Phase IIb multicenter trial of vorinostat in patients with persistent, progressive, or treatment refractory cutaneous T-cell lymphoma. J Clin Oncol. 2007 Jul 20;25(21):3109-15. doi: 10.1200/JCO.2006.10.2434. Epub 2007 Jun 18. PMID 17577020
- [Background] Fantin VR, Loboda A, Paweletz CP, Hendrickson RC, Pierce JW, Roth JA, Li L, Gooden F, Korenchuk S, Hou XS, Harrington EA, Randolph S, Reilly JF, Ware CM, Kadin ME, Frankel SR, Richon VM. Constitutive activation of signal transducers and activators of transcription predicts vorinostat resistance in cutaneous T-cell lymphoma. Cancer Res. 2008 May 15;68(10):3785-94. doi: 10.1158/0008-5472.CAN-07-6091. PMID 18483262
- Available data/document: CSR Snyopsis Links — http://www.merck.com/clinical-trials/policies-perspectives.html